CLINICAL TRIAL: NCT00787800
Title: Reduction And Prevention of Tachyarrhythmias and Shocks Using Reduced Ventricular Pacing With Atrial Algorithms (The RAPTURE Study)
Brief Title: The Use of Dual Chamber ICD With Special Programmed Features to Lower the Risk of Inappropriate Shock
Acronym: RAPTURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Paul A. Friedman, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-003618
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Atrial Fibrillation; Supraventricular Tachycardia
Keywords: Shock prevention; Single vs. Dual Chamber; Reduce ventricular pacing; Atrial Fibrillation; Remote Monitoring; ICD; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual Chamber ICD (Active Comparator): Dual chamber Implantable Cardioverter-Defibrillator (ICD): Atrial therapies and minimized ventricular pacing will be programmed on along with Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) detection and therapies with detection enhancements; remote monitoring set to alert for sustained atrial fibrillation.
  Interventions: Device: Dual Chamber ICD
- Single Chamber ICD (Active Comparator): Single chamber Implantable Cardioverter-Defibrillator: Optimally programmed Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) detection and therapies will be programmed on including use of detection enhancements.
  Interventions: Device: Single Chamber ICD

INTERVENTIONS:
Device: Dual Chamber ICD — Dual Chamber ICD: Atrial therapies and minimized ventricular pacing will be programmed on along with VT/VF detection and therapies with detection enhancements; remote monitoring set to alert for sustained atrial fibrillation Dual Chamber ICD Atrial prevention and termination therapies, Managed Ventricular Pacing (MVP)along with VT/VF detection and therapies for dual chamber device.
  Other Names: Virtuoso DR D154AWG
  Arms: Dual Chamber ICD
Device: Single Chamber ICD — Single Chamber: Optimally programmed VT/VF detection and therapies will be programmed on including use of detection enhancements.
  VT/VF detection and therapies with discrimination criteria for single chamber device.
  Other Names: Virtuoso VR D154VWC
  Arms: Single Chamber ICD

SUMMARY:
The RAPTURE Study will determine whether dual chamber defibrillators with atrial prevention and termination therapies, minimized ventricular pacing, and remote monitoring will reduce the rate of inappropriate shocks and improve quality of life compared to optimally programmed back-up pacing only single chamber ICDs when used for primary prevention of sudden cardiac death

DETAILED DESCRIPTION:
While implantable cardioverter-defibrillator (ICD) therapy has become the gold standard for sudden death prevention in high risk individuals, reduction of device associated morbidity remains a significant problem. Rapidly conducted atrial tachyarrhythmias inappropriately detected as ventricular tachycardia (VT) are the most common cause for inappropriate shocks in ICD recipients, affecting 10 to 40% of patients. Large multicenter trials have shown modest benefits of atrial pacing in preventing atrial fibrillation, however right ventricular (RV) pacing was not limited, thus any favorable effects associated with atrial prevention and treatment may have been offset by the RV pacing. New algorithms to prevent RV pacing are now made available in our current devices. The choice of dual chamber versus single chamber ICD for primary prevention warrants re-assessment of atrial prevention and termination therapies, without the potentially adverse effects of RV pacing.

This Multi Center Pilot study will enroll 100 eligible subjects, 50 to single chamber and 50 to dual chamber ICDs. Patients will be followed for one year.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for ICD for primary prevention according to American Heart Association/American College of Cardiology (AHA/ACC) guidelines who have a clinical indication for ICD implantation for ventricular arrhythmia or sudden death prevention.
* The ability to understand the scope of the study, provide written informed consent, and a willingness to complete all study visits and associated procedures.

Exclusion Criteria:

* Pregnant women
* Age <18 years old
* Inability to provide consent
* On a heart transplant waiting list
* Life expectancy <1 year
* Indication for pacing
* Atrioventricular (AV) node ablation
* Permanent atrial fibrillation or atrial flutter
* Indication for cardiac resynchronization
* Preexisting, separate pacemaker pulse generator that won't be explanted
* Intra-aortic balloon pump or other device
* Inotropic drug (not digitalis) necessary for hemodynamic support
* Chronic serious bacterial infection
* Inability to receive pectoral non-thoracotomy lead ICD
* Inability to program device according to protocol
* History of Out of Hospital Cardiac Arrest (OHCA) or sustained Ventricular Tachycardia as an indication for ICD (secondary prevention indication)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Friedman, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
- Israel (2):
  - Carmel Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan

REFERENCES:
- [Background] Deisenhofer I, Kolb C, Ndrepepa G, Schreieck J, Karch M, Schmieder S, Zrenner B, Schmitt C. Do current dual chamber cardioverter defibrillators have advantages over conventional single chamber cardioverter defibrillators in reducing inappropriate therapies? A randomized, prospective study. J Cardiovasc Electrophysiol. 2001 Feb;12(2):134-42. doi: 10.1046/j.1540-8167.2001.00134.x. PMID 11232608
- [Background] Friedman PA, McClelland RL, Bamlet WR, Acosta H, Kessler D, Munger TM, Kavesh NG, Wood M, Daoud E, Massumi A, Schuger C, Shorofsky S, Wilkoff B, Glikson M. Dual-chamber versus single-chamber detection enhancements for implantable defibrillator rhythm diagnosis: the detect supraventricular tachycardia study. Circulation. 2006 Jun 27;113(25):2871-9. doi: 10.1161/CIRCULATIONAHA.105.594531. Epub 2006 Jun 12. PMID 16769912
- [Background] Theuns DA, Rivero-Ayerza M, Boersma E, Jordaens L. Prevention of inappropriate therapy in implantable defibrillators: A meta-analysis of clinical trials comparing single-chamber and dual-chamber arrhythmia discrimination algorithms. Int J Cardiol. 2008 Apr 25;125(3):352-7. doi: 10.1016/j.ijcard.2007.02.041. Epub 2007 Apr 18. PMID 17445918
- [Background] Sweeney MO, Bank AJ, Nsah E, Koullick M, Zeng QC, Hettrick D, Sheldon T, Lamas GA; Search AV Extension and Managed Ventricular Pacing for Promoting Atrioventricular Conduction (SAVE PACe) Trial. Minimizing ventricular pacing to reduce atrial fibrillation in sinus-node disease. N Engl J Med. 2007 Sep 6;357(10):1000-8. doi: 10.1056/NEJMoa071880. PMID 17804844
- [Background] Friedman PA, Bradley D, Koestler C, Slusser J, Hodge D, Bailey K, Kusumoto F, Munger TM, Militanu A, Glikson M. A prospective randomized trial of single- or dual-chamber implantable cardioverter-defibrillators to minimize inappropriate shock risk in primary sudden cardiac death prevention. Europace. 2014 Oct;16(10):1460-8. doi: 10.1093/europace/euu022. Epub 2014 Jun 13. PMID 24928948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2008 to 2010, patients who were undergoing Implantable Cardioverter-Defibrillators (ICD) device implantation at Mayo Clinic in Rochester, Minnesota and Jacksonville, Florida and at two Israeli medical center sites, Sheba Medical Center in Ramat Gan and Carmel Medical Center in Haifa, were screened for entry into this open-label study.
Groups:
- Dual Chamber ICD: Dual chamber Implantable Cardioverter-Defibrillator (ICD): Atrial therapies and minimized ventricular pacing will be programmed on, along with Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) detection and therapies with detection enhancements; remote monitoring set to alert for sustained atrial fibrillation.
- Single Chamber ICD: Single chamber Implantable Cardioverter-Defibrillator: Optimally programmed VT/VF detection and therapies will be programmed on including use of detection enhancements.
Period: Overall Study
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Started | 50 | 50
Completed | 47 | 43
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dual Chamber ICD: Dual chamber Implantable Cardioverter-Defibrillator (ICD): Atrial therapies and minimized ventricular pacing will be programmed on along with VT/VF detection and therapies with detection enhancements; remote monitoring set to alert for sustained atrial fibrillation.
- Total: Total of all reporting groups
Arm/Group | Dual Chamber ICD | Single Chamber ICD | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Date of birth not obtained for 4 Israeli subjects (treatment arm unknown).
  years | 62.6 (12.4) | 59.9 (14.8) | 61.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 42 | 41 | 83
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
  Israel | 25 | 25 | 50
NYHA Classification [Number; unit: Participants] — New York Heart Association (NYHA) classification of Heart Failure is used to describe the degree of limitation due to heart failure at baseline.
  I. No limitation, II. Limitation with ordinary activity, III. Limitation with less than daily activity, IV. Symptoms at rest, (NA-Not applicable; participants without heart failure)
  Participants
    I- No limitation | 8 | 11 | 19
    II- Limitation with ordinary activity | 24 | 23 | 47
    III-Limitation with less than daily activity | 8 | 10 | 18
    IV-Symptoms at rest | 1 | 0 | 1
    NA-No heart failure | 7 | 5 | 12
    Heart Failure present but NYHA class not recorded | 2 | 1 | 3
LV Ejection Fraction [Mean (Standard Deviation); unit: Percentage of LV blood volume] — Left ventricular Ejection Fraction (LVEF) is a clinical parameter used by cardiologists to describe how well the heart is pumping. LVEF is a calculated measure of the amount of blood pumped out of the lower chamber of the heart during a heartbeat, measured using echocardiography. A normal LVEF ranges from 55-70%. A LVEF of 65, for example, means that 65% of the total amount of blood in the left ventricle is pumped out with each heartbeat. Note: LVEF baseline data is missing for one Israeli subject, arm unknown.
  Percentage of LV blood volume | 30.1 (14.1) | 29.6 (13.3) | 29.9 (13.7)
Co-morbidities [Number; unit: participants] — Participants could have had more than one co-morbidity, therefore the sum total of co-morbid conditions will not equal the total number of participants.
  participants
    Pulmonary Disease | 1 | 7 | 8
    Diabetes | 15 | 18 | 33
    Hypertension | 32 | 26 | 58
    Hyperlipidemia | 34 | 36 | 70
    Stroke | 2 | 3 | 5
    Transient Ischemic Attack | 0 | 3 | 3
    History of Paroxysmal Atrial Fibrillation | 6 | 3 | 9
Cardiac Disease [Number; unit: Participants] — Participants could have more than one concomitant cardiac disease event/diagnosis, therefore the sum total of all cardiac conditions will not equal the total number of participants.
  Participants
    Coronary Artery Disease | 35 | 36 | 71
    Myocardial Infarction | 31 | 35 | 66
    Percutaneous Coronary Intervention | 23 | 27 | 50
    Coronary Artery Bypass Graft | 16 | 20 | 36
    Hypertrophic Cardiomyopathy | 6 | 6 | 12
    Dilated Cardiomyopathy | 13 | 10 | 23
Concomitant Medications [Number; unit: Participants] — Each category lists the number of participants taking each medication.
  Participants
    Beta Blocker | 47 | 44 | 91
    Calcium Channel Blocker | 2 | 3 | 5
    Amiodarone | 1 | 3 | 4
Ventricular Depolarization (QRS) Duration [Mean (Standard Deviation); unit: milliseconds] — Note:QRS baseline data is missing for one Israeli subject. As the heart undergoes depolarization and repolarization, the electrical currents that are generated spread within the heart & throughout the body. This electrical activity can be measured by electrodes placed on the body surface & produce a tracing called an electrocardiogram (ECG, or EKG). The different waves that comprise the ECG represent the sequence of depolarization and repolarization of the atria and ventricles. Certain points on the ECG tracing are assigned letters. The QRS complex represents ventricular depolarization.
  milliseconds | 112.1 (26.3) | 103.9 (18.2) | 108.4 (23.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Inappropriately Shocked by Implantable Cardioverter-Defibrillator (ICD)
Description: An inappropriate shock is defined as a shock delivered by the ICD during a rhythm other than sustained VT/VF (ventricular tachycardia/ventricular fibrillation).
Time Frame: Baseline to 12 months after ICD implantation
Population: Intent to Treat population analyzed.
Measure: Number; unit: Participants
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 50 | 50
Participants | 1 | 1
Statistical Analysis 1: Comparison: Dual Chamber ICD vs Single Chamber ICD; Test type: Superiority or Other; p = 1.0, Log Rank

2. Secondary Outcome: Number of Atrial Tachyarrhythmia Episodes Lasting Over 5 Minutes
Description: Episodes of Atrial Fibrillation (AF) or Atrial Flutter (AFL) greater than 5 minutes duration. A subject may experience multiple episodes.
Time Frame: Baseline to 12 Months
Population: Intent to Treat population analyzed. 37 episodes in 5 subjects (all in dual chamber arm).
Measure: Number; unit: Episodes
Groups:
- Dual Chamber ICD: Dual chamber Implantable Cardioverter-Defibrillator (ICD): Atrial therapies and minimized ventricular pacing will be programmed on, along with VT/VF detection and therapies with detection enhancements; remote monitoring set to alert for sustained atrial fibrillation.
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 50 | 50
Episodes | 37 | 0

3. Secondary Outcome: Number of Appropriate Shocks by ICD
Description: Appropriate shocks are delivered during a sustained Ventricular Tachycardic/Ventricular Fibrillation heart rhythm.
Time Frame: Baseline to 12 Months
Population: Intent to Treat population analyzed.
Measure: Number; unit: Shocks
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 50 | 50
Shocks | 31 | 1
Statistical Analysis 1: Comparison: Dual Chamber ICD vs Single Chamber ICD; Test type: Superiority or Other; p = 0.050, t-test, 2 sided

4. Secondary Outcome: Total Cost of ICD Implantation Procedure
Time Frame: Baseline
Population: Only the 45 subjects enrolled at Mayo Clinic in Rochester, Minnesota were analyzed for ICD implantation costs.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 23 | 22
US Dollars | 16,579 (1,359) | 14,249 (1,421)

5. Secondary Outcome: Number of Subjects With Newly Detected Atrial Tachyarrhythmias
Time Frame: Baseline to 12 months after ICD implantation
Population: Intent to Treat population analyzed.
Measure: Number; unit: Participants
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 50 | 50
Participants | 12 | 0
Statistical Analysis 1: Comparison: Dual Chamber ICD vs Single Chamber ICD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Atrial Fibrillation (AF) Burden
Description: AF burden is defined as the sum of duration of all atrial arrhythmias divided by total observation time, reported as a percentage value.
Time Frame: Implantation through 1 year
Population: Intent to treat analysis population.
Measure: Mean (Standard Deviation); unit: Percentage of atrial arrhythmias per min
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Number analyzed (Participants) | 50 | 50
Percentage of atrial arrhythmias per min | 0.02 (0.07) | 0 (0)

ADVERSE EVENTS:
Time Frame: Implantation of ICD to one year.
Arm/Group | Dual Chamber ICD | Single Chamber ICD
Serious Adverse Events (participants affected / at risk) | 8/50 | 8/50
Other Adverse Events (participants affected / at risk) | 16/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Chamber ICD (N=50) | Single Chamber ICD (N=50)
Death (General disorders) | 0 (0) | 2 (2) — The cause of death for two Israeli subjects was not reported.
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cancer spreading (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Defibrillator Threshold testing could not be done at implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fluid overload (Cardiac disorders) | 0 (0) | 1 (1)
High Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Right ventricular lead replaced (Surgical and medical procedures) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Venous thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Chamber ICD (N=50) | Single Chamber ICD (N=50)
Hematoma/Seroma (Vascular disorders) | 2 (2) | 0 (0)
Infection/Erosion (Infections and infestations) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pneumothorax/Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Phlebitis/Thrombosis/Embolism (Vascular disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident/Transient Ischemic Attack (Vascular disorders) | 1 (1) | 0 (0)
Device dislodgement from ventricle (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Device Oversensing-Atrial (Surgical and medical procedures) | 4 (5) | 0 (0)
Device Oversensing-Ventricle (Surgical and medical procedures) | 3 (3) | 1 (1)
Device Failure to Capture-Atrial (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No